CLINICAL TRIAL: NCT00273091
Title: MODULA-Study: Modul 5 / BEAT HF: Detektion and Registration of Atrial Tachyarrhythmias at Patients With Heart Failure
Brief Title: MODULA Modul 5 BEAT-HF
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Guidant Corporation (Industry)
Responsible Party: jens goetzke, guidant germany a boston scientific company
Other Study IDs: Version vom 10.07.2003
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: ICD with CRT therapy — permanently CRT pacing

SUMMARY:
Detektion and Registration of Atrial Tachyarrhythmias at Patients with Heart Failure; What proportion of patients with CRT-therapy are affected at least temporarily by Atrial Arrhythmia?

DETAILED DESCRIPTION:
How many patients with CRT-therapy are affected at least temporarily by Atrial Arrhythmia in terms of rate, characteristics and severity of atrial rhythm disturbances at patients with CRT-therapy within 12 months after implantation of a CRT-device.

ELIGIBILITY:
Inclusion Criteria:

* patient under CRT-D or CRT-P therapy

Exclusion Criteria:

* patients with permanent Atrial Fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elegible patients comprise the investiagators standard CRT-D population.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2003-08; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of atrial tachycardia in CRT patients | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Burkhard J. Hügl, phd, Principal Investigator — Herzzentrum / Klinik für Kardiologie / Robert-Koch-Allee 9 / 99437 Bad Berka / Germany
Locations (1):
- Herzzentrum / Klinik für Kardiologie / Robert-Koch-Allee 9, Bad Berka, Germany